CLINICAL TRIAL: NCT07178210
Title: Robotic-Enabled Microsurgical Intervention for Neurodegenerative Disease - A Global, Prospective, Early Feasibility Study in Alzheimer's Patients
Brief Title: Robotic-Enabled Microsurgical Intervention for Neurodegenerative Disease
Acronym: REMIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-00157
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Lymphatic Obstruction
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Alzheimer's Disease (Experimental): Patient with confirmed mild to moderate Alzheimer's Disease according to the National Institute of Aging-Alzheimer's Association (NIA-AA) criteria
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — Use of Symani Surgical System for performing microsurgical techniques in the deep cervical lymph nodes.

SUMMARY:
The objective of this investigational device exemption (IDE) study is to evaluate the safety and feasibility of using the Symani System and microsurgical techniques in the deep cervical lymph node (dCLN) region in the setting of mild to moderate Alzheimer's disease and lymphatic abnormalities.

DETAILED DESCRIPTION:
A prospective, multi-center, early feasibility study, designed to evaluate the Symani System's safety and feasibility for performing microsurgical techniques in the dCLN region to improve clearance of neurotoxins, such as amyloid-beta and phosphorylated tau, in patients with confirmed mild to moderate Alzheimer's disease and lymphatic abnormalities in the dCLN region.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 50 or older
2. Patient has confirmed mild to moderate Alzheimer's Disease according to the National Institute of Aging-Alzheimer's Association (NIA-AA) criteria
3. Patient has a positive amyloid PET test and/or a positive CSF t-tau/amyloid-beta-42 test
4. Patient has an MMSE score within the mild to moderate range (21-26 and 10-20)
5. Patient has CDR-SB score within the mild to moderate range; mild is 4.5to 9.0 and moderate is 9.5 to 15.5
6. Patient has confirmed extracranial lymphatic abnormalities in the head and neck region as identified by preoperative imaging
7. Investigator deems the candidate acceptable for lymphatic surgery with a robotic-assisted microsurgical anastomosis in accordance with the Symani System's Instructions for Use (IFU)
8. Patient or their legally authorized representative agrees to participate in the study, return for all required follow-up visits, complete all study procedures, and has willingly provided written informed consent after receiving all information related to the study, its requirements, and the robotic assisted procedure

Exclusion Criteria:

1. Patient (or their legally authorized representative) is unwilling to provide informed consent
2. Patient has suspected dementia of other type, e.g., Lewy body, frontotemporal disorder, vascular, etc.
3. Patient has documented or suspected neurological or intracranial conditions such as cerebrovascular accident, tumors, intracranial space occupying lesions, seizures or other intracranial/neurological conditions that may affect their safety in the study.
4. History of head and neck radiation exposure
5. Patient with severe kidney disease (GFR <30 mL/min/1.73m2)
6. Patient with acute kidney injury
7. Active systemic infection under treatment with intravenous antibiotics
8. Patient has a modified Rankin Score (mRS) of >4
9. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders, previous mental disorders, or other disorders that may significantly affect the data collection or the ability to comply with the protocol per the investigator's discretion
10. Known history of significant bleeding, coagulopathy, or Von Willebrand's disease
11. Patient with an active cancer diagnosis and/or currently receiving treatment for cancer or has received treatment within the past 6 months
12. Patient is currently receiving treatment or has been treated with anti-amyloid-beta monoclonal antibody therapy within the past 3 months
13. Patient has contraindication for MRI or intrathecal administration of gadobutrol
14. Currently enrolled in any other investigational clinical studies that the investigator believes may impact patient safety or study outcomes
15. Patient is ineligible to participate for other reasons in the judgment of the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Device-related serious adverse events at 30-days | The duration of the participants' index procedure through 30-days post index procedure.
  All intraoperative and postoperative device-related serious adverse events (SAEs) will be captured from the start of the index procedure through 30 days post-index procedure for each participant. The device-related SAE rate will be reported at 30 days post-index procedure for all evaluable participants.

SECONDARY OUTCOMES:
Rate of Serious Adverse Events (SAEs) at 6 months | The duration of the participants' index procedure through 6-months post index procedure.
  All intraoperative and postoperative SAEs, regardless of device relatedness, will be captured from the start of the index procedure through 6 months days post-index procedure for each participant. The freedom from SAE rate will be reported at 6 months post-index procedure for all evaluable participants.
Rate of Adverse Events (AEs) at 30 days | The duration of the participants' index procedure through 30-days post index procedure.
  All intraoperative and postoperative AEs, regardless of seriousness or device relatedness, will be captured from the start of the index procedure through 3 months days post-index procedure for each participant. The freedom from AE rate will be reported at 3 months post-index procedure for all evaluable participants.
Anastomosis-Specific Reoperation Rate at 30 Days | The duration of the participants' index procedure through 30-days post index procedure.
  An anastomosis-specific reoperation is defined as a reoperation to revise a robotic anastomosis, which may consist of the addition of stitches, the removal of stitches, or any other form of reoperation directly to robotic anastomoses performed in the index procedure. All anastomosis-specific reoperations will be captured from the end of the index procedure through 30 days post-index procedure for each participant. All anastomosis-specific reoperations will be reviewed by a DSMB Charter. The anastomosis-specific reoperation rate will be reported at 30 days post-index procedure for all evaluable participants.
Change in Amyloid PET Centiloid Value at 6 Months | The duration of the participants' pre-procedure visit through 6-months post index procedure.
  The centiloid (CL) value of an amyloid positron emission tomography (PET) imaging test will be recorded at the patient's pre-procedure visit and at the 6-month follow-up visit.
Change in Plasma Biomarkers at 6 Months: amyloidβ-42 and 40, ptau-217, NfL and GFAP | The duration of the participants' pre-procedure visit through 6-months post index procedure.
  Blood panel testing for amyloidβ-42 and 40, ptau-217, neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP) will be taken at the patient's pre-procedure visit and at the 6-month follow-up visit.
Anastomosis Patency Prior to Closure | The duration of the participants' index procedure.
  Intraoperative patency of the anastomosis should be assessed prior to closure per site standard of care. This information will be captured for each robotic anastomosis performed during the procedure.
Intraoperative Conversion to Manual Approach | The duration of the participants' index procedure.
  The rate of conversion to manual approach will be measured during the index procedure for each participant. This information will be captured for each robotic anastomosis performed during the procedure.